CLINICAL TRIAL: NCT04077879
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP1617 in Healthy Adult Non-Asian and Japanese Subjects Including an Assessment of a Food Effect
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP1617 in Healthy Adult Non-Asian and Japanese Subjects Including Assessment of a Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1617-CL-1001
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: ASP1617; Food Effect; Pharmacokinetics; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single ascending dose of ASP1617 (Experimental): This is composed of 5 sequential cohorts (cohorts 1.1 to 1.5), 6-9 participants for each cohort, consisting of either only non-Asians in cohorts 1.1 and 1.2; or non-Asians plus Japanese in cohorts 1.3, 1.4 and 1.5). Participants in cohorts 1.1, 1.2, 1.3, 1.4 and 1.5 will receive a single dose of 2, 10, 30, 100 and 300 milligrams (mg) ASP1617 capsules respectively under fasting conditions
  Interventions: Drug: ASP1617
- Single ascending dose of Placebo (Placebo Comparator): Participants (2-3 for each cohort, consisting of either only non-Asians in cohorts 1.1 and 1.2; or non-Asians plus Japanese in cohorts 1.3, 1.4 and 1.5) will receive a single dose of matching placebo under fasting conditions.
  Interventions: Drug: Placebo
- Single dose of ASP1617 (Food Effect) (Experimental): Participants (6 Japanese and 3 non-Asian) will receive a single dose of 100 mg ASP1617 with a high-fat meal. Dosing of the Food Effect cohort will commence after having established the safety and tolerability of the dose tested in cohort 1.4.
  Interventions: Drug: ASP1617
- Multiple ascending dose of ASP1617 (Experimental): This is composed of 3 sequential cohorts (cohorts 2.1 to 2.3, 9 participants for each cohort, consisting of only non-Asians in cohort 2.1, or non-Asians plus Japanese in cohorts 2.2 and 2.3). Participants in cohorts 2.1, 2.2 and 2.3 will receive 30, 60 and 110 mg ASP1617 capsules respectively twice daily for 14 consecutive days at the same dose level.
  Based on safety, tolerability and pharmacokinetic data of Part 1, once daily or twice daily dosing will be selected.
  Interventions: Drug: ASP1617
- Multiple ascending dose of Placebo (Placebo Comparator): Participants (3 for each cohort, consisting of either only non-Asians in cohort 2.1, or non-Asians plus Japanese in cohort 2.2 and 2.3) will receive matching Placebo for 14 consecutive days at the same dose level in cohort 2.1 to 2.3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1617 — Oral
  Arms: Multiple ascending dose of ASP1617; Single ascending dose of ASP1617; Single dose of ASP1617 (Food Effect)
Drug: Placebo — Oral
  Arms: Multiple ascending dose of Placebo; Single ascending dose of Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending oral doses of ASP1617 in healthy adult non-Asian and Japanese male and female participants.

This study also evaluate the pharmacokinetics and determine the effect of food on the pharmacokinetics of a single oral dose of ASP1617.

DETAILED DESCRIPTION:
After a screening period of up to 28 days prior to study drug administration, eligible participants will be residential for a single period of 8 days/7 nights in Part 1: single ascending dose, and 21 days/20 nights in Part 2 multiple ascending dose.

ELIGIBILITY:
Inclusion Criteria:

* For cohorts that enroll non-Asian subjects, subject does not have East Asian (China, Hong Kong, Macau, Japan, Mongolia, North Korea, South Korea and Taiwan) ancestries.
* For cohorts that enroll Japanese subjects, subject is first generation Japanese, born in Japan with 4 grandparents of Japanese descent, and must have resided outside of Japan for ≤ 10 years.
* Subject has a body mass index (BMI) range of 18.5 to 32.0 kg/m2, inclusive and weighs at least 50 kg at screening.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Male subject with female partner(s) of child-bearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 30 days after final IP administration.
* Male subject must not donate sperm during the treatment period and for 30 days after final IP administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition, which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP1617 or any components of the formulation used.
* Subject has had previous exposure with ASP1617.
* Subject has any of the liver function tests (alkaline phosphatase [ALP], ALT, AST, gamma glutamyl transferase and TBL) above the upper linit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Subject has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial or fungal infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure (SBP)140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Subject has a mean QTcF of > 430 msec (for male subjects) and > 450 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Subject has used any prescribed or nonprescribed drugs in the 2 weeks prior to first IP administration, except for occasional use of acetaminophen (up to 2 g/day) topical dermatological products, including corticosteroid products, hormonal contraceptives or hormone replacement therapy (HRT).
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening.
* Subject has a history of consuming > 14 units for male subjects or > 7 units for female subjects of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening or the subject tests positive for alcohol at screening or on day -1.
* Subject has used any drugs of abuse within 3 months prior to day -1 or the subject tests positive for drugs of abuse at screening or on day -1.
* Subject has used any inducer of metabolism in the 3 months prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus (HAV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.
* Subject has received any Coronavirus Disease 2019 (COVID-19) vaccines within 14 days prior to first IP administration.
* Subject has received any Coronavirus Disease 2019 (COVID-19) vaccines within 14 days prior to first IP administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) in Part 1 | Up to Day 16
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP) and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
  AE is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
  An AE with onset at any time from first dosing until last scheduled procedure will be classified as a treatment-emergent adverse event (TEAE). A drug-related TEAE is defined as any TEAE with a causal relationship assessed as "yes" by the investigator, or records where the relationship is missing.
Number of participants with laboratory value abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs in Part 1 | Up to Day 16
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with AEs in Part 2 | Up to Day 29
  An AE is any untoward medical occurrence in a subject administered an IP and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.
  AE is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
  An AE with onset at any time from first dosing until last scheduled procedure will be classified as a TEAE. A drug-related TEAE is defined as any TEAE with a causal relationship assessed as "yes" by the investigator, or records where the relationship is missing.
Number of participants with laboratory value abnormalities and/or AEs in Part 2 | Up to Day 29
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or AEs in Part 2 | Up to Day 29
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-ECG abnormalities and/or AEs in Part 2 | Up to Day 29
  Number of participants with potentially clinically significant 12-ECG values.

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics (PK) of ASP1617 in plasma: area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 7
  AUCinf will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1617 in plasma: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to Day 7
  AUClast will be recorded from the PK plasma samples collected.
Part 1: PK of ASP1617 in plasma: maximum concentration (Cmax) | Up to Day 7
  Cmax will be recorded from the PK plasma samples collected.
Part 2 (first dose): PK of ASP1617 in plasma: AUC from the time of dosing to 12 hours (AUC12) | Up to 12 hours
  AUC12 will be recorded from the PK plasma samples collected.
Part 2 (first dose and last dose): PK of ASP1617 in plasma: Cmax | Up to Day 17
  Cmax will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1617 in plasma: AUC during a dosing interval, where tau(τ) is the length of the dosing interval (AUCtau) | Up to Day 17
  AUCtau will be recorded from the PK plasma samples collected.
Part 2 (last dose): PK of ASP1617 in plasma: accumulation ratio calculated using AUC (Rac(AUC)) | Up to Day 17
  Rac(AUC) will be recorded from the PK plasma samples collected.
PK of ASP1617 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to Day 17
  Ctrough will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- California Clinical Trials Medical Group / Parexel, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kojima T, Chen W, Smulders R, Stanhope S, Kowalski D, Heo N, Moy S, Goldston A, Han D, Zhu T. First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ASP1617, a Cathepsin-S Inhibitor, in Healthy Adult Subjects. Clin Transl Sci. 2026 Feb;19(2):e70460. doi: 10.1111/cts.70460. PMID 41577633